CLINICAL TRIAL: NCT06885580
Title: The Effects of Digital Media Privacy Literacy Education on Children's Autonomy, Decision-making and Privacy Awareness
Brief Title: Digital Media Privacy Literacy Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Reyhan Yalcın, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AtaturkU-RY-1
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Student; Digital Health Literacy; Autonomy
Keywords: children; digital privacy literacy; autonomy; decision making; privacy awareness
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Students will be assigned to 2 groups: experimental and control group.
Who Masked: Outcomes Assessor
Masking Description: Data collection tools will be collected by an interviewer independent of the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education (Experimental): Digital privacy literacy training will be provided in 8 sessions over a 12-week period.
  Interventions: Behavioral: Education
- Control (No Intervention): No educational intervention

INTERVENTIONS:
Behavioral: Education — Students will be provided with digital privacy literacy training designed using the puzzle method, which will consist of 8 sessions over a 12-week period.
  Arms: Education

SUMMARY:
The purpose of this randomized controlled experimental study is to evaluate the effects of digital privacy literacy education on children's autonomy, decision-making and privacy awareness.The hypotheses of the study are as follows; H1a: Digital privacy literacy education has an effect on children's autonomy. H1b: Digital privacy literacy education has an effect on children's decision-making.

H1c: Digital privacy literacy education has an effect on children's privacy awareness.

DETAILED DESCRIPTION:
The research will be conducted with 4th grade students (9-12 years old) who are receiving education in a primary school affiliated to Ağrı Provincial Directorate of National Education and who meet the inclusion criteria. Students will be divided into 2 groups as experimental and control groups by simple random method. Digital environment privacy literacy training will be provided to the experimental group, while no training will be provided to the control group. Data will be collected using "Child Information Form", "Autonomy Survey" and "Primary School Students' Privacy Consciousness Scale".

ELIGIBILITY:
Inclusion Criteria

* Being in the 4th grade of primary school
* Not being an inclusive student
* Parent's written consent to participate in the research
* Child's verbal consent to participate in the research

Exclusion Criteria

* Child/parent wants to leave the study at any stage
* Child does not attend the training sessions 2 or more times
* Child does not complete at least one of the pre-test and post-test data collection tools

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Autonomy Survey | 1 weeks
  The survey was developed to determine the level of autonomy of 4th and 5th grade primary school students. The autonomy survey consists of 2 sections. The first section contains 20 items regarding children's decisional autonomy. The second section contains 19 items regarding children's behavioral autonomy. The survey is a four-point Likert-type scale and is scored as never: 1, sometimes: 2, often: 3, always: 4. There are no reverse-coded items in the survey. All items in the survey are collected according to their sections to measure the relevant autonomy. As the total score obtained from the survey increases, the level of autonomy also increases. Researchers found the Cronbach-Alpha internal consistency coefficient of the survey as .84.
  In this study, the first section of the autonomy survey, decisional autonomy, was used. Scores between 20 and 80 are obtained from this section.
Privacy Awareness Scale of Primary School Students | 1 weeks
  It was developed to determine the level of privacy awareness of primary school 3rd and 4th grade students. The scale consists of 4 factors and 16 items. These factors are; Personal Security, Sharing of Personal Information, Social Media Privacy, Parental Control. The scale is a 3-point Likert type and is scored as disagree: 1, undecided: 2, agree: 3. There are 2 reverse items in the scale (items 7 and 13). The score that can be obtained from the scale varies between 16 and 48 points. The sub-factors and total score in the scale are obtained by adding the item scores.
Introductory Information Form | 1 weeks
  The introductory information form, which was created by the researcher by scanning the relevant literature, consists of a total of 9 questions regarding the student's age, gender, mother's education level, father's education level, socioeconomic status, who owns the digital device he/she uses to access the internet, the frequency of use of digital devices, the purpose for which he/she uses the internet, and whether he/she has a social media account.

SECONDARY OUTCOMES:
Autonomy survey | 12 weeks
  The survey was developed to determine the level of autonomy of 4th and 5th grade primary school students. The autonomy survey consists of 2 sections. The first section contains 20 items regarding children's decisional autonomy. The second section contains 19 items regarding children's behavioral autonomy. The survey is a four-point Likert-type scale and is scored as never: 1, sometimes: 2, often: 3, always: 4. There are no reverse-coded items in the survey. All items in the survey are collected according to their sections to measure the relevant autonomy. As the total score obtained from the survey increases, the level of autonomy also increases. Researchers found the Cronbach-Alpha internal consistency coefficient of the survey as .84. In this study, the first section of the autonomy survey, decisional autonomy, was used. Scores between 20 and 80 are obtained from this section.
Privacy Awareness Scale of Primary School Students | 12 weeks
  It was developed to determine the level of privacy awareness of primary school 3rd and 4th grade students. The scale consists of 4 factors and 16 items. These factors are; Personal Security, Sharing of Personal Information, Social Media Privacy, Parental Control. The scale is a 3-point Likert type and is scored as disagree: 1, undecided: 2, agree: 3. There are 2 reverse items in the scale (items 7 and 13). The score that can be obtained from the scale varies between 16 and 48 points. The sub-factors and total score in the scale are obtained by adding the item scores.

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Kadiroğlu, PhD, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No